CLINICAL TRIAL: NCT04840992
Title: A Randomized, Double-blind, Placebo-Controlled Phase I/II Clinical Trial to Evaluate the Safety and Immunogenicity of Ad5-nCoV for Inhalation in Adults 18 Years of Age and Older
Brief Title: Phase I/II Clinical Trial of Recombinant Novel Coronavirus (COVID-19) Vaccine (Adenovirus Type 5 Vector) for Inhalation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CanSino Biologics Inc. (Industry)
Collaborators: Beijing Institute of Biotechnology (Other); Jiangsu Province Centers for Disease Control and Prevention (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: JSVCT092
Record Dates: First submitted 2021-04-08; First posted 2021-04-12 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-10

CONDITIONS: COVID-19
Keywords: COVID-19; Vaccine; Ad5; Safety; Immunogenicity; SARS-CoV-2; Adenovirus Vector; Aerogen Solo
MeSH Terms: conditions — COVID-19; Alzheimer Disease 5 | interventions — Inhalation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (22):
- A1a Phase I low 2 doses (Experimental): Ad5-nCoV containing 0.5E10 vp, 2 doses 56 days apart, Aerogen Solo
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) for Inhalation
- A1b Phase I placebo low 2 doses (Placebo Comparator): Placebo containing 0 vp, 2 doses 56 days apart, Aerogen Solo
  Interventions: Biological: Placebo for Inhalation
- A2a Phase I medium 2 doses (Experimental): Ad5-nCoV containing 1E10 vp, 2 doses 56 days apart, Aerogen Solo
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) for Inhalation
- A2b Phase I placebo medium 2 doses (Placebo Comparator): Placebo containing 0 vp, 2 doses 56 days apart, Aerogen Solo
  Interventions: Biological: Placebo for Inhalation
- A3a Phase I high 2 doses (Experimental): Ad5-nCoV containing 2E10 vp, 2 doses 56 days apart, Aerogen Solo
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) for Inhalation
- A3b Phase I placebo high 2 doses (Placebo Comparator): Placebo containing 0 vp, 2 doses 56 days apart, Aerogen Solo
  Interventions: Biological: Placebo for Inhalation
- A4a Phase I combine 2 doses (Experimental): 1 dose Intramuscular Injection, Ad5-nCoV containing 5E10 vp, 1 dose Aerogen Solo, Ad5-nCoV containing 2E10 vp, 56 days apart
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) for Inhalation; Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector)
- A4b Phase I placebo combine 2 doses (Placebo Comparator): 6 subjects, Placebo containing 0 vp, 1 dose Intramuscular Injection, 1 dose Aerogen Solo, 56 days apart
  Interventions: Biological: Placebo for Inhalation; Biological: Placebo
- A5a Phase I single dose (Experimental): Ad5-nCoV containing 1E10 vp, 1 dose Aerogen Solo
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) for Inhalation
- A5b Phase I placebo single dose (Placebo Comparator): 6 subjects, Placebo containing 0 vp, 1 dose Aerogen Solo
  Interventions: Biological: Placebo for Inhalation
- B1a Phase II low 2 doses (Experimental): Ad5-nCoV containing 0.5E10 vp, 2 doses 56 days apart, Aerogen Solo
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) for Inhalation
- B1b Phase II placebo low 2 doses (18-59) (Placebo Comparator): Placebo containing 0 vp, 2 doses 56 days apart, Aerogen Solo
  Interventions: Biological: Placebo for Inhalation
- B2a Phase II medium 2 doses (Experimental): Ad5-nCoV containing 1E10 vp, 2 doses 56 days apart, Aerogen Solo
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) for Inhalation
- B2b Phase II placebo medium 2 doses (Placebo Comparator): Placebo containing 0 vp, 2 doses 56 days apart, Aerogen Solo
  Interventions: Biological: Placebo for Inhalation
- B3a Phase II high 2 doses (Experimental): Ad5-nCoV containing 2E10 vp, 2 doses 56 days apart, Aerogen Solo
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) for Inhalation
- B3b Phase II placebo high 2 doses (Placebo Comparator): Placebo containing 0 vp, 2 doses 56 days apart, Aerogen Solo
  Interventions: Biological: Placebo for Inhalation
- B4a Phase II combine 2 doses (Experimental): 1 dose Intramuscular Injection, Ad5-nCoV containing 5E10 vp, 1 dose Aerogen Solo, Ad5-nCoV containing 2E10 vp, 56 days apart
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) for Inhalation; Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector)
- B4b Phase II placebo combine 2 doses (Placebo Comparator): Placebo containing 0 vp, 1 dose Intramuscular Injection, 1 dose Aerogen Solo, 56 days apart
  Interventions: Biological: Placebo for Inhalation; Biological: Placebo
- B5a Phase II intramuscular single dose (Experimental): Ad5-nCoV containing 5E10 vp, 1 dose Intramuscular Injection
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector)
- B5b Phase II placebo intramuscular single dose (Placebo Comparator): placebo containing 0 vp, 1 dose Intramuscular Injection
  Interventions: Biological: Placebo
- B6a Phase II Aerogen Solo single dose (Experimental): Ad5-nCoV containing 1E10 vp, 1 dose Aerogen Solo
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) for Inhalation
- B6b Phase II placebo Aerogen Solo single dose (Placebo Comparator): placebo containing 0 vp, 1 dose Aerogen Solo
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector)

INTERVENTIONS:
Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) for Inhalation — Aerogen Solo
  Arms: A1a Phase I low 2 doses; A2a Phase I medium 2 doses; A3a Phase I high 2 doses; A4a Phase I combine 2 doses; A5a Phase I single dose; B1a Phase II low 2 doses; B2a Phase II medium 2 doses; B3a Phase II high 2 doses; B4a Phase II combine 2 doses; B6a Phase II Aerogen Solo single dose
Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) — Intramuscular administration
  Arms: A4a Phase I combine 2 doses; B4a Phase II combine 2 doses; B5a Phase II intramuscular single dose; B6b Phase II placebo Aerogen Solo single dose
Biological: Placebo for Inhalation — Aerogen Solo
  Arms: A1b Phase I placebo low 2 doses; A2b Phase I placebo medium 2 doses; A3b Phase I placebo high 2 doses; A4b Phase I placebo combine 2 doses; A5b Phase I placebo single dose; B1b Phase II placebo low 2 doses (18-59); B2b Phase II placebo medium 2 doses; B3b Phase II placebo high 2 doses; B4b Phase II placebo combine 2 doses
Biological: Placebo — Intramuscular administration
  Arms: A4b Phase I placebo combine 2 doses; B4b Phase II placebo combine 2 doses; B5b Phase II placebo intramuscular single dose

SUMMARY:
This study is a randomized, double-blind, placebo-controlled I/II clinical trial, in order to evaluate the safety and immunogenicity of Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) for Inhalation in adults 18 years of Age and Older.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18 years of age and above at the time of enrollment;
* Able to provide consent to participate in and having signed an Informed Consent Form (ICF);
* Able and willing to complete all the scheduled study procedures during the whole study follow-up period;
* HIV negative;
* No nasal or oral diseases, such as acute rhinitis (sinusitis), allergic rhinitis, oral ulcers, sore throat, etc;
* IgG ang IgM negative for Covid-19;
* Axillary temperature ≤37.0℃;
* No contact history of Covid-19.

Exclusion Criteria:

* Serious cardiovascular diseases, such as arrhythmia, conduction block, myocardial infarction, severe hypertension and uncontrollable medications (on-site measurement: systolic blood pressure ≥160mmHg, diastolic blood pressure ≥100mmHg), etc;
* Abnormal laboratory test indicators which investigator decide to be clinically significant; (Only Phase I volunteers)
* Respiratory rate ≥17 per minute;
* Abnormal lung function such as asthma, chronic obstructive pulmonary disease, pulmonary fibrosis, etc;
* Prior Covid-19 vaccinations;
* Symptoms of upper respiratory track infections;
* Medical or family history of convulsions, epilepsy, encephalopathy, and psychosis disorders;
* History of allergies to any ingredient of Ad5-nCoV, history of serious allergic reactions to any vaccine, history of allergies and immune diseases;
* Acute febrile diseases and infectious diseases;
* Medical history of SARS (SARS-CoV-1);
* Severe chronic diseases or with advanced stage conditions which cannot be controlled smoothly, such as diabetes, thyroid disease, etc;
* Congenital or acquired angioedema/neurological edema;
* Urticaria history within 1 year before receiving the study vaccine;
* Asplenia or functional asplenia;
* Thrombocytopenia or other coagulation disorders (may cause contraindications for intramuscular injection);
* Trypanophobia in intramuscular injection groups;
* History of receiving immunosuppressant therapy (continuous oral or instillation for more than 14 days), anti-allergic therapy, cytotoxic therapy, nebulized corticosteroid therapy in the past 6 months;
* Prior administration of blood products in last 4 months;
* Other vaccination(s) or investigational drugs within 1 month before study onset, or planned use during the study period;
* Prior administration of live attenuated vaccine within 1 month before study onset;
* Prior administration of subunit or inactivated vaccine within 14 days before study onset;
* Current anti-tuberculosis therapy;
* Women who are pregnant or lactating, positive urine pregnancy test or plan to become pregnant during the whole study;
* Any condition that in the opinion of the investigators may interfere with the participants' compliance or evaluation of study objectives or informed consent (i.e. medical, psychological, social or other conditions, etc.) Exclusion criteria for the phase II portion of the study will be detailed in an amended synopsis/study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 840 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-08-09 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Reactions (AR) | 0-14 days after each vaccination
  The occurrence of Adverse Reactions (AR) in all groups
Incidence of Serious Adverse Events (SAE) | Within the first and final vaccination up until 12 months after the final vaccination
  The occurrence of Serious Adverse Events (SAE) in all groups

SECONDARY OUTCOMES:
Incidence of Adverse Events/Reactions (AE/AR) | Within 0-7 days after each vaccination
  The occurence of Adverse Events/Reactions (AE/AR) in all groups
Incidence of Adverse Events/Reactions (AE/AR) | Within 0-28 days after each vaccination
  The occurence of Adverse Events/Reactions (AE/AR) in all groups
Changes in laboratory test indicators | 4 days after each vaccination
  Changes in laboratory test indicators (including white blood cell count, lymphocyte count, etc), and respiratory rate in all groups
GMT of Covid-19 S protein RBD specific antibody | Before the first dose, 28 days after first dose, before the second dose, 14 days after the second dose
  GMT of S protein RBD specific antibody by ELISA
Seroconversion rate of Covid-19 S protein RBD specific antibody | Before the first dose, 28 days after first dose, before the second dose, 14 days after the second dose
  Seroconversion rate of S protein RBD specific antibody by ELISA
GMI of Covid-19 S protein RBD specific antibody | Before the first dose, 28 days after first dose, before the second dose, 14 days after the second dose
  GMI of S protein RBD specific antibody by ELISA
GMT of SARS-CoV-2 neutralizing antibody | Before the first dose, 28 days after the first dose, before the second dose, 14 days after the second dose
  GMT of SARS-CoV-2 neutralizing antibody against pseudovirus
Seroconversion rate of SARS-CoV-2 neutralizing antibody | Before the first dose, 28 days after the first dose, before the second dose, 14 days after the second dose
  Seroconversion rate of SARS-CoV-2 neutralizing antibody against pseudovirus
GMI of SARS-CoV-2 neutralizing antibody | Before the first dose, 28 days after the first dose, before the second dose, 14 days after the second dose
  GMI of SARS-CoV-2 neutralizing antibody against pseudovirus
GMT of SARS-CoV-2 neutralizing antibody | 28 days after the final vaccination
Seroconversion rate of SARS-CoV-2 neutralizing antibody | 28 days after the final vaccination
Cellular immune response | Before the first dose, 14 days after the first dose
  The positive rate of IFN-γ stimulated by S protein ELISpot
Cellular immune response | Before the first dose, 14 days after the first dose
  The positive rate of TNF-α stimulated by S protein ELISpot
Cellular immune response | Before the first dose, 14 days after the first dose
  The positive rate of IL-5 stimulated by S protein ELISpot
Cellular immune response | Before the first dose, 14 days after the first dose
  The positive rate of IL-4 stimulated by S protein ELISpot
Cellular immune response | Before the first dose, 14 days after the first dose
  The positive rate of IL-13 stimulated by S protein ELISpot

CONTACTS AND LOCATIONS:
Overall Officials: Fengcai Zhu, MSD, Principal Investigator — Jiangsu Provincal Center for Disease Control and Prevention
Locations (1):
- Jiangsu Provincal Center for Disease Control and Prevention, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhu Y, Tang R, Li X, Chen X, Wang X, Wang Y, Wang R, Zhu F, Li J. Vaccination with Adenovirus Type 5 Vector-Based COVID-19 Vaccine as the Primary Series in Adults: A Randomized, Double-Blind, Placebo-Controlled Phase 1/2 Clinical Trial. Vaccines (Basel). 2024 Mar 11;12(3):292. doi: 10.3390/vaccines12030292. PMID 38543926
- [Derived] Xia X, Tan ZM, Wan P, Zheng H, Tang R, Chen XQ, Guo XL, Zhu T, Feng JL, Zhong J, Li XL, Zhang ZY, Zhu FC, Li JX. Environmental Impact Assessment for the Use of an Orally Aerosolized Adenovirus Type-5 Vector-Based COVID-19 Vaccine in Randomized Clinical Trials. J Infect Dis. 2023 Sep 15;228(6):715-722. doi: 10.1093/infdis/jiad134. PMID 37202147